CLINICAL TRIAL: NCT01721057
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib (LY3009104) in Patients With Inadequate Response to Conventional Disease-Modifying Antirheumatic Drugs With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: A Study in Moderate to Severe Rheumatoid Arthritis Participants
Acronym: RA-BUILD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14059; I4V-MC-JADX (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-11-01; First posted 2012-11-02 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered orally once daily through Week 24. Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 milligram (mg) orally once daily through Week 24.
  Participants will continue to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
  Interventions: Drug: Placebo; Drug: cDMARD
- Baricitinib 2 mg (Experimental): Baricitinib 2 mg administered orally once daily through Week 24. Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 mg orally once daily through Week 24.
  Participants will continue to take background cDMARD therapy throughout study.
  Interventions: Drug: Baricitinib; Drug: cDMARD
- Baricitinib 4 mg (Experimental): Baricitinib 4 mg administered orally once daily through Week 24. Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 mg orally daily through Week 24.
  Participants will continue to take background cDMARD therapy throughout study.
  Interventions: Drug: Baricitinib; Drug: cDMARD

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Baricitinib — Administered orally
  Other Names: LY 3009104; INCB 028050
  Arms: Baricitinib 2 mg; Baricitinib 4 mg
Drug: cDMARD — Conventional disease-modifying anti-rheumatic drug as a background therapy

SUMMARY:
The purpose of this study is to determine whether baricitinib 4 milligram (mg) once daily (QD) is superior to placebo in the treatment of participants with moderately to severely active Rheumatoid Arthritis (RA) who have had inadequate response to or are intolerant to at least 1 conventional disease-modifying antirheumatic drug (cDMARD)(cDMARD-IR [inadequate response] participants) and who have not received a biologic disease-modifying antirheumatic drug (DMARD).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset Rheumatoid Arthritis (RA) as defined by the American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) 2010 Criteria for the Classification of RA
* Have moderately to severely active RA defined as the presence of at least 6/68 tender joints and at least 6/66 swollen joints
* Have a C-reactive protein (CRP) or high-sensitivity C-reactive protein (hsCRP) measurement ≥ (greater than or equal to) 1.2 times the upper limit of normal (ULN)
* Have had an insufficient response or are intolerant to conventional disease-modifying antirheumatic drugs (cDMARDs) and either:

  * Have had regular use of a cDMARD for at least the 12 weeks prior to study entry with a continuous, nonchanging dose for at least 8 weeks prior to study entry
  * For participants not receiving a cDMARD at the time of entry, the investigator will document in the participant's history that the participant had failed, was unable to tolerate, or had a contraindication to treatment with a cDMARD

Exclusion Criteria:

* Are currently receiving corticosteroids at doses > (greater than)10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of study entry or within 6 weeks of planned randomization
* Have started treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or have been receiving an unstable dosing regimen of NSAIDs within 2 weeks of study entry or within 6 weeks of planned randomization
* Are currently receiving concomitant treatment with methotrexate (MTX), hydroxychloroquine, and sulfasalazine or combination of any 3 cDMARDs
* Have ever received any biologic DMARD
* Have received interferon therapy within 4 weeks prior to study entry or are anticipated to require interferon therapy during the study
* Have received any parenteral corticosteroid administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study
* Have had 3 or more joints injected with intraarticular corticosteroids or hyaluronic acid within 2 weeks prior to study entry or within 6 weeks prior to planned randomization
* Have active fibromyalgia that, in the investigator's opinion, would make it difficult to appropriately assess RA activity for the purposes of this study
* Have a diagnosis of any systemic inflammatory condition other than RA, such as, but not limited to juvenile chronic arthritis,spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, active vasculitis or gout(participants with secondary Sjogren's syndrome are not excluded.)
* Have a diagnosis of Felty's syndrome
* Have had any major surgery within 8 weeks of study entry or will require major surgery during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the participant
* Have experienced any of the following within 12 weeks of study entry: myocardial infarction, unstable ischemic heart disease, stroke, or have New York Heart Association stage IV heart failure
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk when taking investigational product or could interfere with the interpretation of data
* Are largely or wholly incapacitated permitting little or no self care, such as, being bedridden or confined to a wheelchair
* Have an estimated glomerular filtration rate (eGFR) based on the most recent available serum creatinine using the Modification of Diet in Renal Disease (MDRD) method of < (less than) 40 milliliter per minute per 1.73 m^2 (mL/min/1.73 m^2)
* Have a history of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the ULN or the most recent available total bilirubin >/=1.5 times the ULN
* Have a history of, lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years
* Have been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination)
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection
* Have had symptomatic herpes zoster infection within 12 weeks prior to study entry
* Have a history of disseminated/complicated herpes zoster (eg, multidermatomal involvement, ophthalmic zoster, central nervous system involvement, postherpetic neuralgia)
* Are immunocompromised and, in the opinion of the investigator, are at an unacceptable risk for participating in the study
* Have a history of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Have screening laboratory test values, including thyroid-stimulating hormone (TSH), outside the reference range for the population or investigative site that, in the opinion of the investigator, pose an unacceptable risk for the participant's participation in the study
* Have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator or the sponsor, are clinically significant and indicate an unacceptable risk for the participant's participation in the study (eg, Fridericia's corrected QT interval >500 millisecond [msec] for men and >520 msec for women)
* Have symptomatic herpes simplex at the time of study enrollment
* Have evidence of active or latent tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (146):
- United States (48):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Desert, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boulder, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewes, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boynton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naples, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vernon Hills, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freehold, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hartsdale, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyomissing, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cypress, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nassau Bay, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Webster, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesapeake, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kennewick, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Franklin, Wisconsin
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Australia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camperdown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maroochydore, Queensland
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merksem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mons
- Canada (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trois-Rivières, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saskatoon, Saskatchewan
- Croatia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Karlovac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varaždin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hustopeče
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uherské Hradiště
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gommern
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Würzburg
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Békéscsaba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- India (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Attavar, Mangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belagavi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gūrgaon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucknow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prato
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valeggio sul Mincio
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nadarzyn
- Portugal (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Almada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponte de Lima
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Germán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Constanța
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulyanovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl
- Slovakia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Partizánske
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topoľčany
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilbao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villajoyosa
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yong Kung City
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, England
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basingstoke, Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Shields, Tyneside

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] van der Heijde D, Kartman CE, Xie L, Beattie S, Schlichting D, Mo D, Durez P, Tanaka Y, Fleischmann R. Radiographic Progression of Structural Joint Damage Over 5 Years of Baricitinib Treatment in Patients With Rheumatoid Arthritis: Results From RA-BEYOND. J Rheumatol. 2022 Feb;49(2):133-141. doi: 10.3899/jrheum.210346. Epub 2021 Sep 15. PMID 34526397
- [Derived] Wells AF, Jia B, Xie L, Valenzuela GJ, Keystone EC, Li Z, Quebe AK, Griffing K, Otawa S, Haraoui B. Efficacy of Long-Term Treatment with Once-Daily Baricitinib 2 mg in Patients with Active Rheumatoid Arthritis: Post Hoc Analysis of Two 24-Week, Phase III, Randomized, Controlled Studies and One Long-Term Extension Study. Rheumatol Ther. 2021 Jun;8(2):987-1001. doi: 10.1007/s40744-021-00317-9. Epub 2021 May 24. PMID 34028703
- [Derived] Thudium CS, Bay-Jensen AC, Cahya S, Dow ER, Karsdal MA, Koch AE, Zhang W, Benschop RJ. The Janus kinase 1/2 inhibitor baricitinib reduces biomarkers of joint destruction in moderate to severe rheumatoid arthritis. Arthritis Res Ther. 2020 Oct 12;22(1):235. doi: 10.1186/s13075-020-02340-7. PMID 33046136
- [Derived] Emery P, Tanaka Y, Cardillo T, Schlichting D, Rooney T, Beattie S, Helt C, Smolen JS. Temporary interruption of baricitinib: characterization of interruptions and effect on clinical outcomes in patients with rheumatoid arthritis. Arthritis Res Ther. 2020 May 15;22(1):115. doi: 10.1186/s13075-020-02199-8. PMID 32414425
- [Derived] Bingham CO 3rd, Gaich CL, DeLozier AM, Engstrom KD, Naegeli AN, de Bono S, Banerjee P, Taylor PC. Use of daily electronic patient-reported outcome (PRO) diaries in randomized controlled trials for rheumatoid arthritis: rationale and implementation. Trials. 2019 Mar 22;20(1):182. doi: 10.1186/s13063-019-3272-0. PMID 30902094
- [Derived] Combe B, Balsa A, Sarzi-Puttini P, Tony HP, de la Torre I, Rogai V, Durand F, Witt S, Zhong J, Dougados M. Efficacy and safety data based on historical or pre-existing conditions at baseline for patients with active rheumatoid arthritis who were treated with baricitinib. Ann Rheum Dis. 2019 Aug;78(8):1135-1138. doi: 10.1136/annrheumdis-2018-214261. Epub 2019 Mar 6. No abstract available. PMID 30842122
- [Derived] Smolen JS, Genovese MC, Takeuchi T, Hyslop DL, Macias WL, Rooney T, Chen L, Dickson CL, Riddle Camp J, Cardillo TE, Ishii T, Winthrop KL. Safety Profile of Baricitinib in Patients with Active Rheumatoid Arthritis with over 2 Years Median Time in Treatment. J Rheumatol. 2019 Jan;46(1):7-18. doi: 10.3899/jrheum.171361. Epub 2018 Sep 15. PMID 30219772
- [Derived] Tanaka Y, McInnes IB, Taylor PC, Byers NL, Chen L, de Bono S, Issa M, Macias WL, Rogai V, Rooney TP, Schlichting DE, Zuckerman SH, Emery P. Characterization and Changes of Lymphocyte Subsets in Baricitinib-Treated Patients With Rheumatoid Arthritis: An Integrated Analysis. Arthritis Rheumatol. 2018 Dec;70(12):1923-1932. doi: 10.1002/art.40680. Epub 2018 Oct 22. PMID 30058112
- [Derived] Wells AF, Greenwald M, Bradley JD, Alam J, Arora V, Kartman CE. Baricitinib in Patients with Rheumatoid Arthritis and an Inadequate Response to Conventional Disease-Modifying Antirheumatic Drugs in United States and Rest of World: A Subset Analysis. Rheumatol Ther. 2018 Jun;5(1):43-55. doi: 10.1007/s40744-018-0110-x. Epub 2018 Apr 21. PMID 29680881
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520
- [Derived] Emery P, Blanco R, Maldonado Cocco J, Chen YC, Gaich CL, DeLozier AM, de Bono S, Liu J, Rooney T, Chang CH, Dougados M. Patient-reported outcomes from a phase III study of baricitinib in patients with conventional synthetic DMARD-refractory rheumatoid arthritis. RMD Open. 2017 Mar 21;3(1):e000410. doi: 10.1136/rmdopen-2016-000410. eCollection 2017. PMID 28405473
- [Derived] Dougados M, van der Heijde D, Chen YC, Greenwald M, Drescher E, Liu J, Beattie S, Witt S, de la Torre I, Gaich C, Rooney T, Schlichting D, de Bono S, Emery P. Baricitinib in patients with inadequate response or intolerance to conventional synthetic DMARDs: results from the RA-BUILD study. Ann Rheum Dis. 2017 Jan;76(1):88-95. doi: 10.1136/annrheumdis-2016-210094. Epub 2016 Sep 29. PMID 27689735

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who did not respond (nonresponders) to study drug were eligible for rescue treatment beginning at Week 16.
  Nonresponders were defined as lack of improvement of at least 20% in both tender joint count and swollen joint count at both Weeks 14 and 16 compared to baseline.
Groups:
- Placebo: Placebo administered orally (PO) once daily (QD)through Week 24.
  Participants continued to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
- Baricitinib 2 mg: Baricitinib 2 mg PO QD through Week 24.
  Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 4 mg: Baricitinib 4 mg PO QD through Week 24.
  Participants continued to take background cDMARD therapy throughout study.
- Rescue: Baricitinib 4 mg administered PO QD through Week 24. Participants continued to take background cDMARD therapy throughout study.
- Placebo-Follow Up; Baricitinib 2 mg- Follow Up: No study drug received. Participants return for safety follow-up visit 28 days after the last dose of study drug.
- Baricitinib 4 mg- Follow Up: No study drug received. Participants return for safety follow-up visit 28 days after the last dose of study drug.
  Includes participants who were rescued to Baricitinib 4 mg.
Period: Treatment Period
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg | Rescue | Placebo-Follow Up | Baricitinib 2 mg- Follow Up | Baricitinib 4 mg- Follow Up
Started | 228 | 229 | 227 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 228 | 229 | 227 | 0 | 0 | 0 | 0
Rescued | 55 | 21 | 15 | 0 | 0 | 0 | 0
Completed | 200 ("Completers" include rescued participants.) | 210 ("Completers" include rescued participants.) | 204 ("Completers" include rescued participants.) | 0 | 0 | 0 | 0
Not Completed | 28 | 19 | 23 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 5 | 8 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 10 | 12 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Rescue Period
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg | Rescue | Placebo-Follow Up | Baricitinib 2 mg- Follow Up | Baricitinib 4 mg- Follow Up
Started | 0 (Participants who were nonresponders based on tender/swollen joint count entered into rescue group.) | 0 (Participants who were nonresponders based on tender/swollen joint count entered into rescue group.) | 0 (Participants who were nonresponders based on tender/swollen joint count entered into rescue group.) | 91 (Participants who were determined to be nonresponders based on tender/swollen joint count.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 88 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Follow Up
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg | Rescue | Placebo-Follow Up | Baricitinib 2 mg- Follow Up | Baricitinib 4 mg- Follow Up
Started | 0 | 0 | 0 | 0 (Rescued participants who entered post-treatment follow-up are included in Baricitinib 4 mg FollowUp) | 17 (Participants from treatment who entered the post-treatment follow-up period.) | 19 (Participants from treatment who entered the post-treatment follow-up period.) | 22 (Participants from treatment and rescue who entered the post-treatment follow-up period.)
Completed | 0 | 0 | 0 | 0 | 17 | 19 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who received at least 1 dose of the study drug.
Groups:
- Placebo: Placebo administered orally (PO) once daily (QD) through Week 24.
  Participants continued to take background cDMARD therapy throughout study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg | Total
Number analyzed (Participants) | 228 | 229 | 227 | 684
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.5) | 52.2 (12.3) | 51.8 (12.1) | 51.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 184 | 187 | 560
  Male | 39 | 45 | 40 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 17 | 44
  Not Hispanic or Latino | 45 | 43 | 43 | 131
  Unknown or Not Reported | 171 | 171 | 167 | 509
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 9 | 14
  Asian | 60 | 61 | 59 | 180
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 10 | 9 | 9 | 28
  White | 153 | 156 | 148 | 457
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 25 | 21 | 18 | 64
  Australia | 8 | 1 | 6 | 15
  Belgium | 1 | 4 | 6 | 11
  Canada | 10 | 10 | 8 | 28
  Croatia | 0 | 2 | 2 | 4
  Czech Republic | 7 | 5 | 3 | 15
  Germany | 4 | 2 | 3 | 9
  Hungary | 7 | 8 | 5 | 20
  India | 19 | 19 | 20 | 58
  Italy | 3 | 3 | 4 | 10
  Japan | 8 | 6 | 7 | 21
  Korea, Republic of | 6 | 7 | 4 | 17
  Mexico | 3 | 8 | 11 | 22
  Poland | 18 | 13 | 20 | 51
  Portugal | 2 | 2 | 1 | 5
  Romania | 1 | 3 | 2 | 6
  Russian Federation | 4 | 10 | 6 | 20
  Slovakia | 3 | 5 | 3 | 11
  Spain | 14 | 10 | 10 | 34
  Taiwan | 26 | 28 | 28 | 82
  United Kingdom | 1 | 4 | 0 | 5
  United States | 58 | 58 | 60 | 176
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: years] — Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who received at least 1 dose of the study drug and had evaluable baseline data.
  years
    number analyzed (Participants) | 228 | 225 | 225 | 678
    (all) | 7.2 (7.5) | 7.6 (7.6) | 7.7 (7.9) | 7.5 (7.6)
Tender Joint Count of 68 Evaluable Joints [Mean (Standard Deviation); unit: Number of Joints] | 24.3 (15.0) | 23.5 (14.1) | 24.3 (14.0) | 24.0 (14.3)
Swollen Joint Count of 66 Evaluable Joints [Mean (Standard Deviation); unit: Number of Joints] | 13.1 (7.2) | 13.6 (8.7) | 13.5 (6.9) | 13.4 (7.6)
High Sensitivity C-Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: milligram per Liter (mg/L)] | 17.7 (20.4) | 18.2 (21.5) | 14.2 (14.5) | 16.7 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% Improvement (ACR20)
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). "ACR20 Responder" is a participant who has at least 20% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity using visual analog scale (VAS), Health Assessment Questionnaire - Disability Index (HAQ-DI), pain due to arthritis, and high-sensitivity C-reactive protein (hsCRP). Participants with missing responses and participants who discontinue study or drug or are rescued before analysis timepoint are deemed non-responders.
Time Frame: Week 12
Population: Modified Intent-to-Treat (mITT) population: all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using non-responder imputation (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
percentage of participants | 39.5 | 65.9 | 61.7
Statistical Analysis 1: Comparison: Placebo vs Baricitinib 4 mg; Test type: Superiority or Other; p = 0.001, Regression, Logistic

2. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty (0 [without any difficulty], 1 [with some difficulty], 2 [with much difficulty], and 3 [unable to do])when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate the HAQ-DI score, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 12
Population: mITT population: all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified baseline observation carried forward (mBOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo administered orally once daily through Week 24.
  Participants continued to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
- Baricitinib 2 mg: Baricitinib 2 mg administered orally once daily through Week 24.
  Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 4 mg: Baricitinib 4 mg administered orally once daily through Week 24.
  Participants continued to take background cDMARD therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
units on a scale | -0.30 (0.45) | -0.52 (0.59) | -0.52 (0.60)

3. Secondary Outcome: Change From Baseline in the Disease Activity Score Based on a 28-Joint Count and High-sensitivity C-reactive Protein (DAS28-hsCRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP) (milligrams per liter), and Patient's Global Assessment of Disease Activity using visual analog scale (VAS) (participant global VAS). DAS28 was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 12
Population: mITT population: all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mBOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
units on a scale | -1.05 (1.23) | -1.83 (1.22) | -1.91 (1.21)

4. Secondary Outcome: Percentage of Participants Achieving Simplified Disease Activity Index (SDAI) ≤3.3
Description: SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Participant's Global Assessment of Disease Activity using VAS centimeters (cm), and Physician's Global Assessment of Disease Activity using VAS (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity. An index-based definition of remission occurs with an SDAI score ≤3.3.
Time Frame: Week 12
Population: mITT population: all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using NRI.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo administered orally (PO) once daily (QD) through Week 24.
  Participants continued to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
- Baricitinib 2 mg: Baricitinib 2 mg PO QD through week 24.
  Participants will continued to take background cDMARD therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
percentage of participants | 0.9 | 9.2 | 8.8

5. Secondary Outcome: Mean Duration of Morning Joint Stiffness(MJS) in the Prior 7 Days as Collected in Electronic Daily Diaries
Description: Participants reported the duration of their morning joint stiffness (MJS) in hours and minutes into daily electronic diaries. If MJS duration was longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses. The average value across the 7 days preceding each visit is calculated. A decrease in duration of MJS indicated an improvement in the participant's condition.
Time Frame: Week 12
Population: mITT population: all randomized participants who received at least 1 dose of the study drug and had at least 4 entries within any post-baseline 7-day window are included in the analysis.
Measure: Median (95% Confidence Interval); unit: minutes
Groups:
- Placebo: Placebo administered orally once daily through Week 24.
  Participants continued disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 221 | 223 | 222
minutes | 60.0 [50.7 to 76.7] | 44.4 [30.0 to 60.0] | 34.6 [23.7 to 51.4]

6. Secondary Outcome: Mean Severity of Morning Joint Stiffness Numeric Rating Scale (NRS) in the Prior 7 Days as Collected in Electronic Diaries
Description: Participants rated the severity of their MJS by selecting a number from 0 to 10 that best described their overall level of MJS from the time they woke up, where 0 represents "no joint stiffness" and 10 represents "joint stiffness as bad as you can imagine". Participants reported their severity daily in electronic diaries. The average value across the 7 days preceding each visit is calculated. A decrease in severity rating indicated an improvement in the participant's condition.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 221 | 223 | 222
units on a scale | 4.2 (2.3) | 3.5 (2.5) | 3.4 (2.2)

7. Secondary Outcome: Mean Worst Tiredness Numeric Rating Scale (NRS) in the Prior 7 Days as Collected in Electronic Diaries
Description: Participants rated their tiredness by selecting a number from 0 to 10 that best described their level of worst tiredness during the past 24 hours, where 0 represents "no tiredness" and 10 represents "as bad as you can imagine". Participants reported their worst tiredness in daily electronic diaries. The average value across the 7 days preceding each visit is calculated. A decrease in tiredness severity rating indicated an improvement in the participant's condition.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 221 | 223 | 222
units on a scale | 4.5 (2.2) | 4.0 (2.5) | 4.0 (2.3)

8. Secondary Outcome: Mean Worst Joint Pain Numeric Rating Scale (NRS) in the Prior 7 Days as Collected in Electronic Diaries
Description: Participants rated their joint pain by selecting a number from 0 to 10 that best described their worst joint pain during the last 24 hours, where 0 represents "no pain" and 10 represents "pain as bad as you can imagine". Participants reported their worst joint pain in daily electronic diaries. The average value across the 7 days preceding each visit is calculated. A decrease in joint pain severity rating indicated an improvement in the participant's condition.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baricitinib 2 mg: Baricitinib 2 mg PO QD through week 24.
  Participants will continue to take background cDMARD therapy throughout study.
- Baricitinib 4 mg: Baricitinib 4 mg PO QD through week 24.
  Participants will continue to take background cDMARD therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 221 | 223 | 222
units on a scale | 4.7 (2.2) | 3.9 (2.5) | 3.8 (2.2)

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 Responder Index is composite of clinical, laboratory, and functional measures in RA. "ACR50 Responder" is a participant who has at least 50% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria:
  Physician Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP. Participants with missing responses and participants who discontinue study or drug or are rescued before analysis timepoint are deemed non-responders.
Time Frame: Week 12, Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo administered orally once daily through Week 24.
  Participants will continue to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
percentage of participants
  Week 12 | 12.7 | 33.6 | 33.5
  Week 24 | 21.5 | 41.5 | 44.1

10. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 Responder Index is composite of clinical, laboratory, and functional measures in RA. "ACR70 Responder" is a participant who has at least 70% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP. Participants with missing responses and participants who discontinue study or drug or are rescued before analysis timepoint are deemed non-responders.
Time Frame: Week 12, Week 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
percentage of participants
  Week 12 | 3.1 | 17.9 | 18.1
  Week 24 | 7.9 | 25.3 | 24.2

11. Secondary Outcome: Change From Baseline in Measures of Clinical Disease Activity Index (CDAI) Score
Description: • The CDAI is a tool for measurement of disease activity in RA that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity. A negative change from baseline indicates improvement in condition.
Time Frame: Baseline, Week 24
Population: mITT population: all randomized participants who received at least 1 dose of the study drug, with a baseline value and at least 1 post-baseline value. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified last observation carried forward (mLOCF) .
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo administered orally once daily through Week 24.
  . Participants continued to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 218 | 224 | 219
units on a scale | -14.29 (16.04) | -20.99 (14.48) | -23.18 (13.47)

12. Secondary Outcome: Change From Baseline in Measures of Simplified Disease Activity Index (SDAI) Score
Description: The SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Patient's Global Assessment of Disease Activity using visual analog scale (cm), and Physician's Global Assessment of Disease Activity using visual analog scale (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity. The SDAI is expressed as a score on a scale with the minimum score=0 (best) to maximum score=86 (worst). A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: mITT population: all randomized participants who received at least 1 dose of the study drug, with a baseline value and at least 1 post-baseline value. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mLOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baricitinib 4 mg: Baricitinib 4 mg administered orally once daily through Week 24.
  Participants will continue to take background cDMARD therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 218 | 224 | 219
units on a scale | -14.55 (16.37) | -21.87 (14.99) | -23.78 (13.94)

13. Secondary Outcome: Change From Baseline in DAS28-Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: DAS28 consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), Erythrocyte Sedimentation Rate (ESR) (millimeters per hour), and Patient's Global Assessment of Disease Activity. DAS28 was calculated using following formula: DAS28-ESR=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.70*natural log(ESR)+0.014*Patient's Global VAS. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 12
Population: mITT population: all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mLOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 220 | 226 | 221
units on a scale | -1.16 (1.27) | -1.89 (1.23) | -1.97 (1.16)

14. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology European League Against Rheumatism (ACR/EULAR) Remission - Boolean Remission
Description: The ACR/EULAR definitions of RA remission includes a Boolean-based definition. The Boolean-based definition of remission occurs when all 4 of the following criteria are met at the same visit: TJC28 ≤1, SJC28 ≤1, acute phase response using C-reactive protein (milligrams per deciliter) ≤1, Patient's Global Assessment of Disease Activity using VAS (cm) ≤1.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
percentage of participants | 0.4 | 7.0 | 6.6

15. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores.
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale is a brief 13-item, symptom-specific questionnaire that specifically assesses the participant's self-reported severity of fatigue and its impact upon daily activities and functioning. The FACIT-F uses a numeric rating scale of 0 ("Not at all") to 4 ("Very much") for each item to assess fatigue and its impact in the past 7 days. Total scores range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: Baseline, Week 12; Baseline Week 24
Population: mITT population: all randomized participants who received at least 1 dose of the study drug , with a baseline value and at least 1 post-baseline value. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mLOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 216 | 227 | 216
units on a scale
  Week 12 | 7.6 (10.3) | 8.7 (11.1) | 8.8 (10.6)
  Week 24 | 7.8 (11.0) | 9.2 (10.7) | 9.7 (10.8)

16. Secondary Outcome: Change From Baseline in Mental Component Score (MCS), Physical Component Score (PCS) of the Medical Outcomes Study 36-Item Short Form Health Survey Version 2 Acute (SF-36v2 Acute)
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (mental [MCS] and physical [PCS]). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baricitinib 4 mg: Baricitinib 4 mg PO QD through week 24.
  Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 mg orally daily through Week 24.
  Participants will continue to take background cDMARD therapy throughout study.
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 218 | 229 | 219
units on a scale
  Week 12, MCS | 3.3 (10.6) | 3.6 (10.5) | 3.3 (11.0)
  Week 24, MCS | 2.7 (11.5) | 3.0 (10.4) | 3.3 (11.3)
  Week 12, PCS | 4.1 (7.3) | 7.7 (8.5) | 7.0 (8.3)
  Week 24, PCS | 4.9 (8.0) | 8.5 (9.0) | 8.6 (9.0)

17. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores
Description: European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. One component consists of a descriptive system of the respondent's health comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state.
Time Frame: Baseline Week 12; Baseline Week 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 216 | 227 | 216
units on a scale
  Index Score (US Algorithm) Week 12 | 0.054 (0.155) | 0.117 (0.151) | 0.109 (0.165)
  Index Score (US Algorithm) Week 24 | 0.051 (0.149) | 0.113 (0.172) | 0.129 (0.173)
  Index Score (UK Algorithm) Week 12 | 0.074 (0.230) | 0.167 (0.221) | 0.159 (0.237)
  Index Score (UK Algorithm) Week 24 | 0.075 (0.218) | 0.162 (0.254) | 0.185 (0.250)

18. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores (Self-Perceived Health)
Description: A second component of the EQ-5D-5L is a self-perceived health score which is assessed using a VAS that ranges from 0 to 100 millimeter (mm), where 0 indicates the worst health you can imagine and 100 indicates the best health you can imagine.
Time Frame: Baseline Week 12; Baseline Week 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 216 | 227 | 216
mm
  Self-Perceived Health, Week 12 | 5.7 (23.8) | 13.4 (21.8) | 11.5 (25.2)
  Self-Perceived Health, Week 24 | 8.4 (25.1) | 13.1 (25.8) | 10.4 (28.8)

19. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) Scores
Description: The Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. It contains 6 items covering overall work productivity (health), overall work productivity (symptom), impairment of regular activities (health), and impairment of regular activities (symptom). Scores are calculated as impairment percentages. The WPAI-RA yields four types of scores: Absenteeism (work time missed), Presenteeism (impairment at work), Work productivity loss (overall work impairment), and Activity impairment.
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: mITT population: all randomized participants who received at least 1 dose of the study drug. Change from baseline includes participants with a baseline value and an observed value at the time point being summarized.
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Placebo | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 228 | 229 | 227
percentage of impairment
  Absenteeism Week 12: number analyzed (Participants) | 73 | 72 | 69
  Absenteeism Week 12 | 2.6 (23.5) | -6.3 (26.5) | 2.5 (24.7)
  Absenteeism Week 24: number analyzed (Participants) | 44 | 62 | 56
  Absenteeism Week 24 | -2.1 (13.9) | -3.8 (28.2) | 4.0 (27.2)
  Presenteeism Week 12: number analyzed (Participants) | 71 | 69 | 66
  Presenteeism Week 12 | -8 (26) | -17 (25) | -15 (27)
  Presenteeism Week 24: number analyzed (Participants) | 44 | 61 | 53
  Presenteeism Week 24 | -17 (26) | -20 (23) | -17 (21)
  Work Productivity Loss Week 12: number analyzed (Participants) | 71 | 69 | 66
  Work Productivity Loss Week 12 | -4.2 (27.7) | -17.6 (30.4) | -9.9 (23.7)
  Work Producivity Loss Week 24: number analyzed (Participants) | 44 | 61 | 53
  Work Producivity Loss Week 24 | -15.9 (26.1) | -19.6 (25.0) | -14.3 (23.0)
  Activity Impairment Week 12: number analyzed (Participants) | 206 | 222 | 213
  Activity Impairment Week 12 | -13 (25) | -19 (27) | -19 (25)
  Activity Impairment Week 24: number analyzed (Participants) | 141 | 187 | 187
  Activity Impairment Week 24 | -18 (27) | -23 (28) | -21 (27)

20. Secondary Outcome: Population Pharmacokinetics (PK): Maximum Concentration at Steady State of Dosing (Cmax,ss) of LY3009104
Time Frame: Week 0: 30 and 90 minutes postdose; Week 8: 1 hour postdose; Week 12, Week 20 and Week 24:predose
Population: All randomized participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 246 | 245
nanogram per milliliter (ng/mL) | 70.2 (26.2) | 138 (25.7)

21. Secondary Outcome: Population PK: Maximum Concentration at Steady State of Dosing (AUC,ss) of LY3009104
Time Frame: Week 0: 30 and 90 minutes postdose; Week 8: 1 hour postdose; Week 12, Week 20 and Week 24; predose
Population: All randomized participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per mL per hour (ng/mL*h)
Arm/Group | Baricitinib 2 mg | Baricitinib 4 mg
Number analyzed (Participants) | 246 | 245
nanograms per mL per hour (ng/mL*h) | 637 (44.5) | 1210 (47)

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo-Treatment Period: Placebo administered orally once daily through Week 24.
  Participants continued to take background conventional disease-modifying antirheumatic drug (cDMARD) therapy throughout study.
- Baricitinib 2 Mg-Treatment Period: Baricitinib 2 mg administered orally once daily through Week 24.
  Participants continued to take background cDMARD therapy throughout study.
- Baricitinib 4 Mg-Treatment Period: Baricitinib 4 mg administered orally once daily through Week 24.
  Participants continued to take background cDMARD therapy throughout study.
Arm/Group | Placebo-Treatment Period | Baricitinib 2 Mg-Treatment Period | Baricitinib 4 Mg-Treatment Period | Rescue | Placebo-Follow Up | Baricitinib 2 mg- Follow Up | Baricitinib 4 mg- Follow Up
Serious Adverse Events (participants affected / at risk) | 13/228 | 6/229 | 12/227 | 1/91 | 1/17 | 0/19 | 1/22
Other Adverse Events (participants affected / at risk) | 105/228 | 108/229 | 127/227 | 21/91 | 2/17 | 0/19 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Treatment Period (N=228) | Baricitinib 2 Mg-Treatment Period (N=229) | Baricitinib 4 Mg-Treatment Period (N=227) | Rescue (N=91) | Placebo-Follow Up (N=17) | Baricitinib 2 mg- Follow Up (N=19) | Baricitinib 4 mg- Follow Up (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo-Treatment Period (N=228) | Baricitinib 2 Mg-Treatment Period (N=229) | Baricitinib 4 Mg-Treatment Period (N=227) | Rescue (N=91) | Placebo-Follow Up (N=17) | Baricitinib 2 mg- Follow Up (N=19) | Baricitinib 4 mg- Follow Up (N=22)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6) | 4 (4) | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3) | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 5 (5) | 4 (4) | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 (4) | 7 (7) | 5 (5) | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 10 (11) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5) | 2 (2) | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 5 (6) | 3 (3) | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 (9) | 7 (7) | 5 (5) | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 (5) | 7 (7) | 4 (4) | 2 (2) | 0 | 0 | 0
Fatigue (General disorders) | 5 (5) | 2 (3) | 5 (5) | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 6 (6) | 3 (3) | 3 (3) | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 (2) | 1 (1) | 5 (7) | 0 | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 11 (12) | 6 (7) | 7 (8) | 2 (2) | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4) | 9 (9) | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 18 (19) | 10 (10) | 18 (22) | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 8 (8) | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 3 (3) | 4 (4) | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 18 (19) | 14 (16) | 24 (26) | 2 (2) | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 (5) | 12 (13) | 9 (9) | 3 (3) | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 (3) | 5 (6) | 5 (6) | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 (2) | 3 (3) | 6 (7) | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 8 (8) | 15 (17) | 0 | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 9 (9) | 4 (4) | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 6 (6) | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (8) | 6 (6) | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (9) | 5 (5) | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 (4) | 3 (3) | 7 (9) | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 (10) | 15 (17) | 9 (10) | 3 (3) | 0 | 0 | 0
Depression (Psychiatric disorders) | 7 (7) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0/39 (0) | 0/45 (0) | 1/40 (1) | 0/13 (0) | 0/6 (0) | 0/4 (0) | 0/3 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/189 (0) | 0/184 (0) | 0/187 (0) | 0/78 (0) | 1/11 (1) | 0/15 (0) | 0/19 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 9 (11) | 9 (10) | 0 | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 9 (9) | 3 (3) | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 6 (6) | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 10 (10) | 6 (6) | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days